CLINICAL TRIAL: NCT01107951
Title: Low-dose Rituximab and High-dose Dexamethasone as First Line Treatment for Adult Patients With Immune Thrombocytopenic Purpura.
Brief Title: Low-dose Rituximab and High-dose Dexamethasone as First Line Treatment for ITP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Medical doctor, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rituximab in PTI 001
Record Dates: First submitted 2010-04-09; First posted 2010-04-21 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Rituximab; Dexamethasone; Low-dose; ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab -dexamethasone (Other): only one arm receive four doses weekly rituximab and four dosis daily dexamethasona
  Interventions: Drug: Rituximab and dexamethasone

INTERVENTIONS:
Drug: Rituximab and dexamethasone — Rituximab 100mg IV days 1,8,15,22.
  Dexamethasone 40mg PO days 1-4 (four days)
  Other Names: Mabthera

SUMMARY:
The purpose of this study is to determine the response rate and response duration with the combination of low-dose rituximab and high-dose dexamethasone in the treatment of adult immune thrombocytopenic purpura.

DETAILED DESCRIPTION:
ITP is an autoimmune disorder characterized by formation of autoantibodies against platelet antigens leading platelet destruction and bleeding. Corticosteroids increase the platelet count in about 80 percent of patients.However, many patients have a relapse when the dose of corticosteroid is reduced. Debilitating side effects are common in patients who require long-term corticosteroid therapy to maintain the platelet count. Rituximab, a chimeric anti-CD20 monoclonal antibody, has been shown to be effectively raise the platelet count in some patients with ITP and there is clinical and biological evidence to suggest that, if given early, rituximab may prevent ITP relapses. Rituximab 375 mg/m2 weekly for four weeks has significant activity in patients with immune thrombocytopenia. Furthermore, using lower dose rituximab the level of B-cell depletion and the response rates appear similar to those previously observed with standard dosages in a population of ITP.

The purpose of this study is to determine the response rate and response duration with the combination of low-dose rituximab (100mg IV days 1,8, 15 and 22) and high-dose dexamethasone (40mg PO days 1,2,3,4) in untreated adult patients immune thrombocytopenic purpura.

A complete platelet response is defined as an increase in platelet counts to >150×109/L on two consecutive occasions. A partial response is defined as an increase in the platelet count to between 50 and 150×109/L on two consecutive occasions, 1 week apart. Duration of response is considered from the day of the initial infusion to the first time of relapse (platelet count <30×109/L)or to time of analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed immune thrombocytopenic purpura (ITP) Platelet count less than 30,000/mm3 on two occasions. Platelets >30000/mm3 with bleeding.
* Normal to increased numbers of megakaryocytes on bone marrow examination in patients ≥ 60 years
* Subject is ≥ 18 years
* Subject has signed and dated written informed consent.
* No sepsis or fever
* No active infection requiring therapy
* No active chronic viral infection
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion Criteria:

* Performance status above or equal to 2.
* Previous treatment with rituximab
* Immunosuppressive treatment within the last month
* Previous splenectomy
* Presence of malignant haematological disease
* Connective tissue disease
* Autoimmune hemolytic anemia
* Pregnancy and lactation
* Not willing to participate in the study.
* Expected survival of < 2 years
* Known intolerance to murine antibodies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-04; Primary Completion 2010-04 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with sustained response after 6 months | 6 months
  Number of patients with partial and complete response after 6 months.

SECONDARY OUTCOMES:
Number of patients with complete response at month 6 | month 6
  Number of patients with platelet count at least 150x109/L, 6 months after therapy
Bleeding | month 6
  Number of patients with bleeding complication after therapy

CONTACTS AND LOCATIONS:
Overall Officials: David Gomez-Almaguer, MD, Principal Investigator — Hospital Universitario
Locations (1):
- Hospital Universitario Dr. Jose E Gonzalez UANL, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Andersen JC. Response of resistant idiopathic thrombocytopenic purpura to pulsed high-dose dexamethasone therapy. N Engl J Med. 1994 Jun 2;330(22):1560-4. doi: 10.1056/NEJM199406023302203. PMID 8177245
- [Background] Cheng Y, Wong RS, Soo YO, Chui CH, Lau FY, Chan NP, Wong WS, Cheng G. Initial treatment of immune thrombocytopenic purpura with high-dose dexamethasone. N Engl J Med. 2003 Aug 28;349(9):831-6. doi: 10.1056/NEJMoa030254. PMID 12944568
- [Background] Zaja F, Battista ML, Pirrotta MT, Palmieri S, Montagna M, Vianelli N, Marin L, Cavallin M, Bocchia M, Defina M, Ippoliti M, Ferrara F, Patriarca F, Avanzini MA, Regazzi M, Baccarani M, Isola M, Soldano F, Fanin R. Lower dose rituximab is active in adults patients with idiopathic thrombocytopenic purpura. Haematologica. 2008 Jun;93(6):930-3. doi: 10.3324/haematol.12206. Epub 2008 Apr 9. PMID 18403395